CLINICAL TRIAL: NCT05222594
Title: Computational Neuroscience of Language Processing in the Human Brain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Principal Investigator, Robert Mark Richardson, Director, Functional Neurosurgery, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020P001989
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Language; Epilepsy
Keywords: language; computational neuroscience; epilepsy
MeSH Terms: conditions — Language; Epilepsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epileptic participants undergoing intracranial monitoring (Other): Patients with pharmaco-resistant epilepsy undergoing intracranial monitoring involving the left cerebral hemisphere.
  Interventions: Other: Behavioral tasks during intracranial monitoring

INTERVENTIONS:
Other: Behavioral tasks during intracranial monitoring — Participants will listen to sentences and stories while neural data are recorded through electrodes placed for clinical purposes.

SUMMARY:
Language is a signature human cognitive skill, but the precise computations that support language understanding remain unknown. This study aims to combine high-quality human neural data obtained through intracranial recordings with advances in computational modeling of human cognition to shed light on the construction and understanding of speech.

DETAILED DESCRIPTION:
The neural architecture of language is the foundation for the highest form of human interaction. Prior work has identified a network of frontal and temporal brain areas that selectively support language processing, but the precise computations that underlie our ability to extract meaning from sequences of words have remained unknown. The standard approaches in human cognitive neuroscience lack the spatial and temporal resolution necessary for precise comparisons to computational models. To bridge this gap in knowledge, neural responses to language stimuli will be collected from epileptic patients undergoing intracranial monitoring. Overall, these data will be used to identify cortical maps of different linguistic manipulations and to better understand properties of the human language network.

ELIGIBILITY:
Inclusion Criteria:

* clinical indications to proceed with intracranial monitoring involving the left cerebral hemisphere, as determined by a multidisciplinary epilepsy surgery team
* the ability to comply with test directions and provide informed consent
* between ages 18 - 85

Exclusion Criteria:

* inability to understand or perform the task outlined in the protocol, or who are unwilling or unable to participate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-02 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Cortical maps of linguistic responses | Throughout intracranial monitoring period, up to approximately 10 days
  By using sEEG intracranial recordings of the brain, EEG power in frequency bands will reflect cortical maps of responses to different linguistic manipulations, informing the functional organization of the human language system. Power is measured in arbitrary units; higher power reflects greater activity at the investigated frequency.
Neural time-courses during naturalistic language comprehension | Throughout intracranial monitoring period, up to approximately 10 days
  Time-courses of neural response to language across diverse parts of the language network. These data will be used to predict across-time variation in response strength from the properties of linguistic input.
Brain scores for diverse artificial neural network (ANN) language models | Throughout intracranial monitoring period, up to approximately 10 days
  Human neural data will be compared to ANN language models to test how well these models predict human responses to language and why. There are no minimum or maximum scores. Higher values mean better model predictivity (i.e., a better match between model representations and neural responses).

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blank I, Balewski Z, Mahowald K, Fedorenko E. Syntactic processing is distributed across the language system. Neuroimage. 2016 Feb 15;127:307-323. doi: 10.1016/j.neuroimage.2015.11.069. Epub 2015 Dec 5. PMID 26666896
- [Background] Blank IA, Fedorenko E. No evidence for differences among language regions in their temporal receptive windows. Neuroimage. 2020 Oct 1;219:116925. doi: 10.1016/j.neuroimage.2020.116925. Epub 2020 May 11. PMID 32407994
- [Background] Fedorenko E, Behr MK, Kanwisher N. Functional specificity for high-level linguistic processing in the human brain. Proc Natl Acad Sci U S A. 2011 Sep 27;108(39):16428-33. doi: 10.1073/pnas.1112937108. Epub 2011 Sep 1. PMID 21885736
- [Background] Fedorenko E, Blank IA. Broca's Area Is Not a Natural Kind. Trends Cogn Sci. 2020 Apr;24(4):270-284. doi: 10.1016/j.tics.2020.01.001. Epub 2020 Feb 20. PMID 32160565
- [Background] Fedorenko E, Duncan J, Kanwisher N. Language-selective and domain-general regions lie side by side within Broca's area. Curr Biol. 2012 Nov 6;22(21):2059-62. doi: 10.1016/j.cub.2012.09.011. Epub 2012 Oct 11. PMID 23063434
- [Background] Fedorenko E, Hsieh PJ, Nieto-Castanon A, Whitfield-Gabrieli S, Kanwisher N. New method for fMRI investigations of language: defining ROIs functionally in individual subjects. J Neurophysiol. 2010 Aug;104(2):1177-94. doi: 10.1152/jn.00032.2010. Epub 2010 Apr 21. PMID 20410363
- [Background] Fedorenko E, Nieto-Castanon A, Kanwisher N. Lexical and syntactic representations in the brain: an fMRI investigation with multi-voxel pattern analyses. Neuropsychologia. 2012 Mar;50(4):499-513. doi: 10.1016/j.neuropsychologia.2011.09.014. Epub 2011 Sep 17. PMID 21945850
- [Background] Fedorenko E, Scott TL, Brunner P, Coon WG, Pritchett B, Schalk G, Kanwisher N. Neural correlate of the construction of sentence meaning. Proc Natl Acad Sci U S A. 2016 Oct 11;113(41):E6256-E6262. doi: 10.1073/pnas.1612132113. Epub 2016 Sep 26. PMID 27671642
- [Background] Mollica F, Siegelman M, Diachek E, Piantadosi ST, Mineroff Z, Futrell R, Kean H, Qian P, Fedorenko E. Composition is the Core Driver of the Language-selective Network. Neurobiol Lang (Camb). 2020 Mar 1;1(1):104-134. doi: 10.1162/nol_a_00005. eCollection 2020. PMID 36794007
- [Background] Nieto-Castanon A, Fedorenko E. Subject-specific functional localizers increase sensitivity and functional resolution of multi-subject analyses. Neuroimage. 2012 Nov 15;63(3):1646-69. doi: 10.1016/j.neuroimage.2012.06.065. Epub 2012 Jul 8. PMID 22784644
- [Background] Norman-Haignere S, Kanwisher NG, McDermott JH. Distinct Cortical Pathways for Music and Speech Revealed by Hypothesis-Free Voxel Decomposition. Neuron. 2015 Dec 16;88(6):1281-1296. doi: 10.1016/j.neuron.2015.11.035. PMID 26687225
- [Background] Pereira F, Lou B, Pritchett B, Ritter S, Gershman SJ, Kanwisher N, Botvinick M, Fedorenko E. Toward a universal decoder of linguistic meaning from brain activation. Nat Commun. 2018 Mar 6;9(1):963. doi: 10.1038/s41467-018-03068-4. PMID 29511192
- [Background] Shain C, Blank IA, van Schijndel M, Schuler W, Fedorenko E. fMRI reveals language-specific predictive coding during naturalistic sentence comprehension. Neuropsychologia. 2020 Feb 17;138:107307. doi: 10.1016/j.neuropsychologia.2019.107307. Epub 2019 Dec 24. PMID 31874149
- [Background] Siegelman M, Blank IA, Mineroff Z, Fedorenko E. An Attempt to Conceptually Replicate the Dissociation between Syntax and Semantics during Sentence Comprehension. Neuroscience. 2019 Aug 10;413:219-229. doi: 10.1016/j.neuroscience.2019.06.003. Epub 2019 Jun 11. PMID 31200104